CLINICAL TRIAL: NCT02188524
Title: The Effect of Training Older Adults in Tai Chi and Compensatory Stepping on Balance Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Dr. Stephen Perry, Professor, Wilfrid Laurier University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM_TCFP
Record Dates: First submitted 2014-05-28; First posted 2014-07-11 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Accidental Falls
Keywords: balance, exercise, compensatory stepping, tai chi
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): No exercise program
- Exercise Group (Experimental): exercise program
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Tai Chi and Compensatory Stepping
  Arms: Exercise Group

SUMMARY:
For the duration of 10 weeks, participants will be asked to maintain their current levels of physical activity and to take part in three testing sessions over the course of 10 weeks. Objective and subjective measurements will be obtained at (week 0), at midpoint (week 5) and after the intervention terminates (week 10). The objective measurements will be taken by inserting pressure sensors directly into the shoe and recording the centre of pressure. Markers will be attached to the surface of the body on the shoulders, feet and belly button and video recording will be used to assess the movement of the centre of mass. The first task requires individuals to stand in one spot with their eyes open, and then eyes closed. Secondly, standing in one place, upon an auditory cue, arms will be lifted to the sky as fast as possible. Lastly, participants will walk around a set of chairs while music plays and when the music stops, this is a cue to stop walking. The Timed-Up-and-Go test requires participants to rise from a seated position, walk 3 meters, turn and return to their original seated position. The Berg Balance Scale requires the completion of a 14 task sequence which evaluates balance ability during seated, and various standing positions as well as transitioning movements. The other measurements taken are collected via a questionnaire about balance confidence level. Upon arrival, participants are required to report whether they have experienced a fall since the last class attended and if yes, a follow-up questionnaire is also required to gain information about the nature of the fall.

DETAILED DESCRIPTION:
The main purpose of my research is to explore the benefits of a 10 week Tai Chi and compensatory stepping training program on balance control among older adults by examining static and dynamic postural responses to perturbations before (0 weeks), at midpoint (5 weeks) and after the intervention (10 weeks). This Tai Chi and compensatory stepping program will be compared to a control group that will not participate in any physical activity for 10 weeks, but will be offered the chance to partake in a fall prevention program after the 10 weeks of testing has been completed. The program will be administered twice weekly for thirty minutes each by experienced instructors at a community location (Lab at WLU). The Tai Chi/compensatory stepping group will engage in 50 minutes of Tai Chi exercise followed by 10 minutes of controlled manual perturbations administered for compensatory stepping training. The control group will not be participating in the Tai Chi and compensatory stepping training during the initial 10 weeks of testing, but will be offered the chance to participate in either the SMART fall prevention program, or given other resources for participation in a fall prevention exercise program. Testing for both groups will take place at baseline (week 0), midpoint (week 5) and post-intervention (week 10). We will be assessing balance control by administering the Berg Balance Scale (attached), the Timed-Up-and-Go Test and tracking the variability, minimum and maximum displacements of the centre of pressure (COP), centre of mass (COM) and maximum and minimum displacement between the COM and COP as an indication of instability. The Activities-Specific Balance Confidence Scale questionnaire (attached) will also be administered as an indication of balance confidence. Tighter regulation of COP and COM and as well as a small displacement between the 2 values indicates greater balance control. COP, COM and COP/COM relationship will be measured during three balance tasks. Participants will have pressure insoles directly inserted into their shoes, markers attached with tape to record movement velocity and change in position. For testing, participants will be required to complete 3 tasks. The first is made up of two parts that measure static balance. Participants will stand in one place with their eyes open for 3 trials for 30 seconds each and then they will be asked to repeat the same standing with their eyes closed. The second task is a measure of static balance in response to a self -perturbation, where participants will raise their arms at a high velocity to the sky to offset balance in response to an unexpected auditory cue. The third task will require participants to walk in a circle around a set of chairs and perturb their balance by terminating gait upon an unexpected auditory cue.

ELIGIBILITY:
Inclusion Criteria:

- age 65+

Exclusion Criteria:

* paralysis
* epilepsy
* cerebral palsy
* multiple sclerosis
* Parkinson's disease
* stroke
* any other neurological disorder
* diabetes
* vision problem other than corrective glasses
* cataract surgery
* a balance or coordination problem
* an inner ear disorder
* hearing problems
* constant ringing in your ears
* ear surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Center of mass - Center of pressure difference | 0,5,10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Perry, PhD, Principal Investigator — Wilfrid Laurier University
Locations (1):
- Biomechanics Lab, Waterloo, Ontario, Canada